CLINICAL TRIAL: NCT05179369
Title: Enhancing Perinatal Care Support to Improve Maternal Mortality Disparities
Brief Title: Well-Mama Community Doula Navigator Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Woman's Hospital, Louisiana (Other); Rutgers University (Other); Cook County Health & Hospitals System (Other)
Responsible Party: Principal Investigator, Melissa Simon, Vice Chair of Research, Professor of Obstetrics and Gynecology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MD016280
Record Dates: First submitted 2021-12-02; First posted 2022-01-05 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Hybrid Type 1 randomized effectiveness-implementation trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants randomized to standard care will be offered prenatal and postpartum care in accordance with site-specific procedures based on AAP and ACOG Guidelines for Perinatal Care. The initial intake appointment, involving a comprehensive visit with physical exam, medical and psychosocial history, laboratory testing, and education would optimally occur in the 1st trimester. Subsequent prenatal visits, per ACOG, is monthly for the first 28 weeks, biweekly for weeks 28-36, and weekly after 36 weeks. More frequent visits may be offered to women at high risk. In addition, some sites may offer supports such as nutritional counseling, childbirth education, and case management. A comprehensive postpartum care visit would typically occur within the first 6 weeks of birth, involving a physical examination, lab tests, and immunizations.
- Standard Care with Well-Mama Intervention (Experimental): Participants will receive standard perinatal care plus the Well Mama intervention, including the Well Mama Checklist, assistance from a Community Doula Navigator, and virtual support groups.
  Interventions: Behavioral: Standard Care with Well-Mama Intervention

INTERVENTIONS:
Behavioral: Standard Care with Well-Mama Intervention — The intervention involves: (1) a Well-Mama checklist on 5 topic areas aligned with leading causes of MM and SMM: (a) mental health/depression; (b) cardiovascular symptoms; (c) safety (e.g., guns at home and intimate partner violence); (d) opioid/substance abuse; and (e) social support, self-agency, and well-being; and (2) Community Doula Navigators (CDNs) who will: (a) conduct biweekly check-ins with pregnant and postpartum women using the Well-Mama List and make appropriate referrals to providers and other resources following check-ins; (b) attend select patient visits; (c) lead virtual pregnancy & postpartum support groups; and (d) provide labor support.
  Arms: Standard Care with Well-Mama Intervention

SUMMARY:
This study will develop and test an intervention, called the Well-Mama intervention, which includes the use of a checklist by Community Doula Navigators to support pregnant women. Participants will be randomized to either receive standard perinatal care or standard perinatal care plus the Well-Mama intervention.

DETAILED DESCRIPTION:
Black, Indigenous, and People of Color (BIPOC) women experience profound maternal health disparities in the US, including rising rates of maternal mortality and severe maternal morbidity. This study will develop a Well-Mama intervention for pregnant and postpartum BIPOC women, centered around Community Doula Navigators conducting in-person and telehealth check-ins on 5 priority areas (mental health, cardiovascular symptoms, safety, opioid/substance abuse, and social support), supplemented with virtual support groups and labor support. The investigators will conduct a randomized trial to test whether the Well-Mama intervention increases BIPOC women's receipt of prenatal and postpartum care.

ELIGIBILITY:
Inclusion Criteria:

1) Pregnant individuals that are age 15-49 years; (2) uninsured or have public insurance (i.e., Medicaid); (3) singleton pregnancy <32 weeks gestation; and (4) not cognitively impaired

Exclusion Criteria:

Already receiving/enrolled in another perinatal care program beyond standard care, such as group prenatal care, maternity home, or employing their own doula

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 576 (Estimated)
Dates: Start 2023-05-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Recommended Perinatal Care Components Received | Baseline through 1 year postpartum
  The primary outcome will be a composite proportion of perinatal care components across three domains, including prenatal care, postpartum care, and social determinants of health content compared between participants in the intervention and control arms.

SECONDARY OUTCOMES:
Level of patient engagement in healthcare management | Baseline through 1 year postpartum
  Patients will complete surveys to measure their level of engagement in their healthcare management .
Level of self-efficacy for dealing with stressful situations | Baseline through 1 year postpartum
  Patients will complete surveys to measure their level of self-efficacy for dealing with stressful situations.
Level of trust in health care system | Baseline through 1 year postpartum
  Patients will complete surveys to measure their level of trust with the health care system.
Rate of experiences of racism and discrimination | Baseline through 1 year postpartum
  Patients will complete surveys to measure their perceived experiences of racism and discrimination while getting health care.
Number of participants with low birth weight newborns | Baseline through 1 year postpartum
  Medical record data extraction will include the number of participants with low birth weight newborns.
Number of participants with NICU admissions | Baseline through 1 year postpartum
  Medical record data extraction will include the number of participants with deliveries resulting in NICU admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa A Simon, MD, MPH, Principal Investigator — Center for Health Equity Transformation Northwestern University
Locations (2):
- United States (2):
  - Woman's Hospital, Baton Rouge, Louisiana
  - University Hospital, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: No